CLINICAL TRIAL: NCT04722653
Title: Investigation of Safety, Tolerability and Pharmacokinetic Properties of Single Subcutaneous Doses of NNC0194-0499 in Japanese and Non-Asian Male Subjects
Brief Title: A Research Study Looking at How the Medicine NNC0194-0499 Behaves in Japanese and Non-Asian Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9500-4663; U1111-1255-1392 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: The present trial is split into two parts reflecting the two trial populations: Japanese subjects and non-Asian subjects. For the Japanese part, it is designed as a randomised, placebo-controlled, double-blinded within cohorts, parallel group, single-dose trial. The non-Asian part is run in parallel to the Japanese part in an open design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The non-Asian part is run in parallel to the Japanese part in an open design. The Japanese part is double-blinded. Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NN0194-0499 (Experimental): Japanese participants will be randomised 3:1 to receive either a single dose of NNC0194-0499 or placebo, Asian participants will only receive NNC0194-0499. There will be 3 cohorts with escalating dose levels. There should be at least 4 days between dose administration of the last participant in a dose level cohort and dose administration of the first participant in the following dose level cohort.
  Interventions: Drug: NNC0194-0499
- Placebo (Placebo Comparator): Japanese participants will be randomised 3:1 to receive either a single dose of NNC0194-0499 or placebo.
  Interventions: Drug: Placebo (NNC0194-0499 )

INTERVENTIONS:
Drug: NNC0194-0499 — 1 single dose administered subcutaneously (s.c. - under the skin)
  Arms: NN0194-0499
Drug: Placebo (NNC0194-0499 ) — 1 single dose administered subcutaneously (s.c. - under the skin).
  Arms: Placebo

SUMMARY:
This study looks at how a new medicine called NNC0194-0499 works in the body of Japanese men and non-Asian men.

Japanese participants will either get NNC0194-0499 or placebo - which treatment participants get is decided by chance. Non-Asian participants will get NNC0194-0499.

Participants will get 1 or 2 injections of the study medicine. It will be injected with a needle into a skin fold on the stomach.

The study will last for a maximum of 66 days. Participants will have 8 scheduled visits with the study doctor. For 1 of the visits participants will stay at the clinic for 6 days (5 nights).

The study includes blood sampling. Participants will not be able to take part in the study if the study doctor thinks there is a risk for participants health.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 20-55 years (both inclusive) at the time of signing informed consent
* For Japanese subjects only, both parents of Japanese descent. For non-Asian subjects only, both parents of non-Asian descent
* Body mass index (BMI) between 23.0 and 34.9 kg/m^2 (both inclusive)
* Body weight greater than or equal to 60 kg

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Subjects aged above or equal to 40 years with an estimated 10-year atherosclerotic cardiovascular disease risk (as described in the American College of Cardiology and the American Heart Association Prevention Guideline) greater than or equal to 5 percentage

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From Day 1 (pre-dose) until completion of the post-treatment period at follow-up (Day 36)
  Count of events

SECONDARY OUTCOMES:
AUC0-∞, SD: The area under the NNC0194-0499 serum concentration-time curve from time 0 to infinity after a single s.c.(subcutaneous) administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  h·nmol/L
AUC0-tz, SD: The area under the NNC0194-0499 serum concentration-time curve from time 0 to the time of the last quantifiable sample after a single s.c. administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  h·nmol/L
AUC0-168h, SD: The area under the NNC0194-0499 serum concentration-time curve from time 0 to 168 hours after a single s.c. administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  h·nmol/L
Cmax, SD: Maximum concentration of NNC0194-0499 in serum after a single s.c. administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  nmol/L
tmax, SD: Time from dose administration to maximum serum concentration of NNC0194-0499 after a single s.c. administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Hours
t½, SD: Terminal half-life of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Hours
CL/FSD: Apparent total serum clearance of NNC0194-0499 | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  L/h
Vz/FSD: Apparent volume of distribution of NNC0194-0499 in the terminal phase | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  L
MRTSD: The mean residence time of NNC0194-0499 after a single s.c. administration | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Dahl K, Friedrichsen MH, Ribel-Madsen R, Hansen JS, Clausen JO, Axelsen M, Palle MS, Lippert SL, Bjorkdahl O, Toubro S, Key C, Andersen B. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Novel Long-Acting FGF21 Analog Zalfermin. Clin Transl Sci. 2025 Dec;18(12):e70435. doi: 10.1111/cts.70435. PMID 41351276